CLINICAL TRIAL: NCT00000760
Title: A Randomized Study of Activity, Safety, and Tolerance of Oral Ro 24-7429 (Tat Antagonist) in Patients With HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Purpose: Treatment
Other Study IDs: ACTG 213; NV14224A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Didanosine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; Gene Products, tat
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ro 24-7429; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Ro 24-7429
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To study the anti-HIV activity of the various doses of Ro 24-7429 monotherapy based on virologic and immunologic endpoints. To study the safety and tolerance of Ro 24-7429. To explore relationships between exposure to Ro 24-7429 and its metabolites and antiviral activity and drug toxicity. To determine a safe, tolerable, and active dose regimen of Ro 24-7429, and to make preliminary observations of Ro 24-7429 in combination with another antiretroviral nucleoside.

The HIV genome contains a number of genes that regulate viral replication. Control of the activity of these genes and their encoded proteins represents a potential target for development of new antiretroviral drugs. The tat (transactivator of transcription of HIV) antagonist Ro 24-7429 is the first compound for clinical testing that utilizes this approach for therapy of HIV infection.

DETAILED DESCRIPTION:
The HIV genome contains a number of genes that regulate viral replication. Control of the activity of these genes and their encoded proteins represents a potential target for development of new antiretroviral drugs. The tat (transactivator of transcription of HIV) antagonist Ro 24-7429 is the first compound for clinical testing that utilizes this approach for therapy of HIV infection.

Ninety-six patients (four treatment arms of 24 patients each) are randomized to receive oral Ro 24-7429 at 1 of 3 doses or nucleoside control (either zidovudine or didanosine). The study will be blinded only for the arms receiving Ro 24-7429. Treatment continues for 12 weeks. After 12 weeks, patients on the nucleoside control arm receive the highest tolerated dose of Ro 24-7429 in addition to their nucleoside.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for P. carinii pneumonia, TB, and mucocutaneous candidiasis.
* Methadone maintenance.
* Hormonal contraceptives.

Patients must have:

* HIV-1 seropositivity.
* CD4 count 50 - 500 cells/mm3.
* Life expectancy of at least 24 weeks.
* Stable weight (+/- 2 kg) by 28 days prior to study entry (by history).

NOTE:

* At least 50 percent of patients must be p24 antigen positive (>= 50 pg/ml).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known or suspected hypersensitivity to benzodiazepines.
* Presence of any malignancy other than basal cell carcinoma or limited cutaneous Kaposi's sarcoma (defined as no more than five lesions with no mucosal involvement).
* Ongoing diarrhea, defined as more than 2 liquid stools per day.
* History, physical exam, or laboratory results consistent with a subclinical AIDS-defining opportunistic infection.
* Grade 2 or greater signs and symptoms of AIDS Dementia Complex.
* Evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, dermatologic, or allergic disease.

Concurrent Medication:

Excluded:

* Chronic suppressive therapy for CMV, MAI, toxoplasmosis, cryptococcosis, cryptosporidiosis, coccidioidomycosis, and histoplasmosis.
* ddC, ddI, AZT (except for control groups) or other experimental antiretrovirals or immunomodulating agents.
* Other medications excluded from the study.

Patients with the following prior conditions are excluded:

* History of serious adverse reactions to benzodiazepines.
* History of intolerance to AZT at 600 mg/day or less or ddI at 400 mg/day or less.
* History of unexplained fever, defined as a temperature of 38.5 deg C or greater with or without night sweats for more than 7 of the past 28 days.

Prior Medication:

Excluded:

* Benzodiazepines within 14 days prior to study entry.

Active drug or alcohol abuse that would interfere with study compliance.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96

CONTACTS AND LOCATIONS:
Overall Officials: Richman DD, Study Chair; Haubrich R, Study Chair
Locations (4):
- United States (4):
  - UCSD, San Diego, California
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Case Western Reserve Univ, Cleveland, Ohio

REFERENCES:
- [Background] Haubrich RH, Flexner C, Lederman MM, Hirsch M, Pettinelli CP, Ginsberg R, Lietman P, Hamzeh FM, Spector SA, Richman DD. A randomized trial of the activity and safety of Ro 24-7429 (Tat antagonist) versus nucleoside for human immunodeficiency virus infection. The AIDS Clinical Trials Group 213 Team. J Infect Dis. 1995 Nov;172(5):1246-52. doi: 10.1093/infdis/172.5.1246. PMID 7594660
- [Background] Haubrich RH. A randomized study of safety, tolerance, pharmacokinetics, and activity of oral Ro 24-7429 (TAT antagonist) in patients with HIV infection. The ACTG 213 Team. Int Conf AIDS. 1993 Jun 6-11;9(1):69 (abstract no WS-B26-5)
- [Background] Lathey JL, Marschner IC, Kabat B, Spector SA. Deterioration of detectable human immunodeficiency virus serum p24 antigen in samples stored for batch testing. J Clin Microbiol. 1997 Mar;35(3):631-5. doi: 10.1128/jcm.35.3.631-635.1997. PMID 9041402